CLINICAL TRIAL: NCT06744179
Title: Understanding the Post-intervention TB Sequelae in Patients After Completion of Standard TB Treatment
Brief Title: Post TB Sequelae Study
Status: Enrolling by invitation | Type: Observational
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: PR-24005
Record Dates: First submitted 2024-10-06; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Echocardiography; Diagnostic Imaging; Blood Cell Count; Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Exposed to pulmonary TB and Not exposed to pulmonary TB: we will enroll a group of individuals exposed to TB who have completed standard TB treatment (e.g., 6-9 months of anti-TB therapy). Simultaneously, we will recruit matched individuals without a history of TB from the same population to form the unexposed group. We will recruit post TB patients and age and sex-matched TB unexposed participants in a 1:1 ratio. We will enrol the unexposed group to compare post-TB sequelae data of study TB patients with that of a local non-TB population. Consequently, we will enrol 210 adult pulmonary TB cases and 90 child TB cases. Similarly, 210 adults and 90 children without TB disease will be included as the unexposed group.
  Interventions: Diagnostic Test: echocardiography, chest x-ray, full blood count , SGPT, lipid profile, HbA1C, AQ20 questionnaire, mmRC dyspnoea scale, Duke activity status index, COPD assessment test, Age and stage questionnaire

INTERVENTIONS:
Diagnostic Test: echocardiography, chest x-ray, full blood count , SGPT, lipid profile, HbA1C, AQ20 questionnaire, mmRC dyspnoea scale, Duke activity status index, COPD assessment test, Age and stage questionnaire — Participants from both exposed and non-exposed groups will be assessed using different standardized questionnaire and a number of investigations to identify any cardiac and pulmonary complications over time. Individuals will be matched for age and sex to ensure comparability. This study aims to evaluate these complications and analyze any significant differences between the groups over the defined follow-up period.

SUMMARY:
The goal of this prospective cohort study is to learn about the long-term health effects of tuberculosis (TB) in children, adolescents, and adults who have completed standard TB treatment in Bangladesh. The study aims to track the evolution of pulmonary and cardiac sequelae within the first two years after TB treatment completion.

The main question it aims to answer is:

Does completing TB treatment result in long-term pulmonary or cardiac health issues (post-TB lung disease, PTLD) in patients compared to those without TB? Additionally, how does this impact children's growth, radiological patterns, and overall quality of life?

Participants who have completed anti-TB treatment for the first episode of pulmonary TB and non-TB participants (age- and sex-matched controls) will be followed for two years. The study will take place at multiple sites in Dhaka, including icddr,b Tuberculosis Screening & Treatment Centers (TBSTC) and Dhaka Shishu Hospital. TB patients and controls will be recruited from Dhaka and surrounding areas.

Over a two-year period, participants will be followed at five key points: within 5-7 days of treatment completion (T0), at 6 months (T1), 12 months (T2), 18 months (T3), and 24 months (T4). Data collection will involve comprehensive clinical evaluations, pulmonary and cardiovascular examinations, laboratory tests, and diagnostic imaging such as chest X-rays, ECGs, and pulmonary function tests.

The study will address several key outcomes, including:

The prevalence and incidence of post-TB lung disease and cardiac sequelae Weight gain and growth in children post-treatment Radiological and ECG patterns post-treatment Mental health and quality of life following TB recovery Associations between demographic, social, and lifestyle factors and post-TB sequelae Through this observational study, researchers hope to contribute valuable insights into the long-term health challenges faced by TB survivors, particularly among children, for whom such data is currently lacking.

DETAILED DESCRIPTION:
Understanding the Post-Intervention TB Sequelae in Patients After Completion of Standard TB Treatment

Introduction:

Tuberculosis (TB) is a chronic infectious disease caused by *Mycobacterium tuberculosis*. It primarily affects the lungs, though it can also involve other tissues. Despite remarkable advances in TB treatment, survivors face substantial health challenges. These include residual lung damage, persistent respiratory symptoms, cardiovascular complications, and even increased mortality risks. This protocol outlines a comprehensive longitudinal cohort study to investigate post-TB sequelae-a critical and under-researched area-focusing on the long-term pulmonary and cardiac health outcomes of TB survivors.

Bangladesh is one of the high TB-burden countries globally, with an incidence rate of 221 cases per 100,000 population and a TB mortality rate of 24 per 100,000 population. Approximately 80% of TB cases in the country are pulmonary TB. The significant burden of TB in Bangladesh underscores the importance of investigating its long-term sequelae to guide health policies and improve patient care.

This study aims to fill critical knowledge gaps, particularly concerning pediatric post-TB health outcomes, by evaluating a cohort of individuals who have completed TB treatment and comparing them with non-TB-exposed counterparts. The study will also assess quality of life, growth in children, and associated mental health outcomes over two years.

Study Rationale:

Post-TB disease, often referred to as post-TB sequelae, includes chronic conditions resulting from TB's impact on the lungs and cardiovascular systems. These sequelae persist despite microbiological cure and have long-term implications on health and quality of life. The following points highlight the rationale for this research:

1. Global Burden: An estimated 10.5 million individuals globally are TB survivors. Evidence suggests that post-TB survivors face a three-fold increased risk of mortality compared to the general population, often due to cardiovascular or respiratory diseases.
2. Knowledge Gaps: While substantial evidence exists on active TB management, little is known about long-term health outcomes post-treatment, particularly in children.
3. Clinical Challenges: Post-TB patients often present with structural and functional lung abnormalities, including fibrosis, bronchiectasis, and chronic airflow obstruction, alongside increased cardiovascular risks such as myocardial infarction.
4. Public Health Implications: Understanding the prevalence, risk factors, and progression of post-TB sequelae is vital for shaping health interventions and policies.

Objectives:

Primary Objective:

To determine the prevalence and incidence of post-TB pulmonary and cardiac sequelae within two years of TB treatment completion among children, adolescents, and adults compared to non-TB populations.

Specific Objectives:

1. Evaluate the incidence of post-TB lung disease (PTLD) within two years of treatment completion.
2. Assess the development of post-TB cardiovascular disease (PTCD) over the same period.
3. Determine case fatality rates among post-TB patients compared to non-TB participants.
4. Identify factors contributing to PTLD and PTCD.
5. Assess growth patterns, including weight gain and linear growth, in pediatric participants.
6. Evaluate quality of life, functional abilities, and mental health in individuals with post-TB sequelae.

Study Design:

Overview This is a prospective, longitudinal cohort study designed to follow TB-exposed and non-TB-exposed populations for two years. The study will enroll participants across different age groups from multiple clinical sites in Dhaka, Bangladesh, including icddr,b and Dhaka Shishu Hospital.

Population:

Participants will be categorized into two cohorts:

1. TB-Exposed Cohort: Individuals who have successfully completed anti-TB treatment.
2. Non-TB Cohort: Age- and sex-matched individuals without TB exposure.

Eligibility Criteria:

Inclusion criteria for TB exposed group

1. Children and adolescents aged 6 months to 15 years; and participants aged >15 years and above.
2. Successful completion of anti-TB treatment for the first episode of pulmonary TB and or pleural TB, with cure or completion as defined by the NTP.
3. Residing within Dhaka city and be willing to come for follow-up visits.(21)
4. Provide consent for participation to the study.

Exclusion criteria

1. Past TB disease or anti-TB treatment within last 6 months.
2. Tuberculous meningitis, and isolated other extra-pulmonary TB (i.e no concomitant pulmonary TB, or pleural TB), multidrug resistant TB.
3. Participants getting immunosuppressive therapy or other chemotherapy for malignancy.
4. Pre-existing mental illness. Participants with preexisting mental illness will be identified based on documented prescriptions or medical records provided by a qualified physician.
5. Participants with known congenital heart disease, ischemic heart disease, cystic fibrosis. These participants will be identified based on documented prescriptions or medical records provided by a qualified physician.
6. Heavy smoker who consumes more than 20 pieces of cigarettes per day or ≥20 more pack-year.

Inclusion criteria for TB unexposed group We will recruit age and sex-matched participants who do not have exposure to TB to compare post-TB sequelae data of study TB patients with that of a local non-TB population. Subjects will be either recruited from the same or neighbouring households of the study TB patients, or from the TBSTCs who will be visiting the centers for TB testing and do not have a TB diagnosis.

Exclusion Criteria for TB unexposed group:

1. Patient will be excluded if any two symptoms or signs suggestive of TB is present according to the national guidelines for the management of TB in children and adult.
2. Past TB disease or anti-TB treatment.
3. Any current or past (chronic) respiratory infection or disease.

   * Documented pneumonia, bronchiolitis, bronchitis in last 3 weeks.
   * Documented asthma, COPD, heart failure diagnosed by medical personnel
   * Documented general wheezing in chest (last 2 years)
   * Self-reported breathing difficulties during mild exercise, or at night. Heavy smoker who consumes more than 20 pieces per day or ≥20 more pack-year.

(**TB symptoms in adolescent and adult:

1. Persistent cough for two weeks or more, with or without production of sputum and despite the administration of a broad spectrum antibiotic.
2. Respiratory symptoms: shortness of breath, chest pain, coughing up of blood.
3. General symptoms: loss of weight, loss of appetite, fever, night sweats.
4. Signs and symptoms of extra-pulmonary TB as listed below

   * TB lymphadenitis: swelling of lymph nodes
   * Pleural effusion: fever, chest pain, shortness of breath
   * TB arthritis: pain and swelling of joints
   * TB of the spine: radiological findings with or without loss of function
   * Meningitis: headache, fever, stiffness of neck and subsequent mental confusion.)

(**TB symptoms in children :

1. Persistent, non-remitting cough for >2 weeks not responding to conventional antibiotics (amoxicillin, co-trimoxazole or cephalosporins) and/or bronchodilators. And/or
2. Persistent documented fever (>380 C/100.40 F) >2 weeks after common cases such as typhoid, malaria or pneumonia have been excluded. And/or
3. Documented weight loss or not gaining weight during the past 3 months (especially if not responding to de-worming together with food and/or micronutrient supplementation) OR severe malnutrition. And/or
4. Fatigue, reduced playfulness, decreased activity.)

Study Procedures:

Patients complying with the eligibility criteria and consenting for participating in the study will be enrolled in the study and will be allocated a unique study ID number.

* Participants will be enrolled within 5-7 days of TB treatment completion.
* Study visits will be conducted at a follow-up clinic at icddr,b at five time points: after treatment completion or cure as defined by NTP (T0), at 6 months (T1), 12 months (T2), 18 months (T3), and 24 months (T4) after enrollment, with a ±1-week window period.
* Baseline data will be collected at the cure or completion of pulmonary TB. All data of prognostic importance, including demographic and social information, as well as lifestyle factors such as smoking and solid fuel sources (e.g., firewood, crop waste, and dung), will be collected. Data on medical history, underlying comorbidities, anthropometric measurements, clinical, laboratory, imaging, and treatment details will be collected using a standard case report form. Information on existing cardiopulmonary diagnoses will be obtained from health records.
* A detailed clinical examination including measurement of vital signs, blood pressure, pulse oximetry, anthropometric measurements, pulmonary, and cardiovascular system examination will be performed by trained research physicians at each follow-up visit. Participants have to stay 1-3 hours per visit at follow-up clinic for this purpose.
* The study team is composed of a qualified pulmonologist and a cardiologist. Consequently, should any cardiopulmonary complications be identified during the study, our expert consultant will offer appropriate management. Additionally, in the event of identifying any mental health issues, we will refer the patient to a psychiatrist for the necessary management.
* Data on health care seeking including unscheduled visit to healthcare provider and hospitalization, TB retreatment will be determined from participant-held health records during the study period. Additionally, we will collect all-cause mortality data from medically certified or registered death records. The WHO verbal autopsy tool will be utilized to document deaths occurring in community settings that are not medically certified or registered.
* Sputum (induced sputum for children) will be collected for Xpert MTB/RIF® and or smear microscopy if indicated.
* Laboratory assessment: We will collect 5 ml of blood through venipuncture to conduct laboratory assays for lipid profile, HbA1C, and capillary blood glucose using a glucometer for children and adolescent. Other tests such as, a complete blood count (CBC), serum alanine transaminase (ALT), serum creatinine will be done if necessary. Additionally, we will perform an electrocardiogram (ECG) and a pulmonary function test. A chest x-ray will be conducted during enrolment after the completion of treatment. Additional tests, such as fasting blood sugar and glycated hemoglobin, will be carried out as needed, especially if the baseline capillary blood glucose (CBG) is high. A high-resolution computed tomography (HRCT) of the chest will be performed if the chest X-ray at T0 time point is abnormal. Additionally, an echocardiogram will be performed in a subset of population.

Follow-Up Visits:

Participants will undergo detailed evaluations at the following time points: T1 (6 months), T2 (12 months), T3 (18 months), and T4 (24 months). Assessments include:

1. Physical Examinations: Comprehensive cardiopulmonary assessments.
2. Imaging: Chest X-rays and HRCT (if indicated).
3. Mental Health Evaluations: PHQ-9 and GAD-7 questionnaires.
4. Growth Assessments: Weight, height, BMI, and mid-upper arm circumference (MUAC) for children.

Data Collection:

Tools:

* Case Report Forms (CRFs): Data will be captured using RedCap®, a secure web-based application.
* Questionnaires: Standardized tools such as the St. George's Respiratory Questionnaire, Airways Questionnaire 20 (AQ20), CAAT Chronic Airway Assessment Test, modified Medical Research Council (mMRC) scale, Duke Activity Status Index (DASI), Patient health (PHQ-9) , The Generalized Anxiety Disorder 7 (GAD-7) tool, Insomnia Severity Index (ISI), Ages and Stages Questionnaires (ASQ), Quality of life questionnaires (PedsQL V.4.0), etc.

Laboratory Tests: Comprehensive blood work and pulmonary function tests.

Quality Control:

Data quality will be ensured through range checks, logical consistency checks, and periodic audits. Confidentiality will be maintained by re-identifying data and restricting access to authorized personnel.

Outcome Measures

Primary Outcomes:

1. Prevalence of PTLD (e.g., chronic cough, dyspnea, abnormal spirometry).
2. Incidence of post-TB cardiac abnormalities (e.g., arrhythmias, heart failure).

Secondary Outcomes:

1. Linear growth rates and weight gain in pediatric participants.
2. Radiological and ECG changes over two years.
3. Mental health status and quality of life.
4. Mortality rates and causes.

Statistical Analysis

Descriptive Statistics:

* Categorical variables: Frequency (%).
* Continuous variables: Mean (SD) or median (IQR).

Inferential Statistics:

1. Bivariate Analysis:

   * Chi-square tests for categorical variables.
   * T-tests or Mann-Whitney U tests for continuous variables.
2. Multivariate Analysis:

   * Mixed-effect models for repeated measures.
   * Cox proportional hazards models for time-to-event data.
3. Survival Analysis:

   * Kaplan-Meier curves for time-to-develop PTLD or PTCD.
   * Log-rank tests for comparing survival curves.

Ethical Considerations Risk Mitigation

* Minimal physical risks associated with diagnostic tests.
* Confidentiality maintained through secure data management.

Benefits:

* Close monitoring of participants for health complications.
* Insights into long-term management of post-TB health outcomes.

Informed Consent:

Participants will provide written informed consent after receiving detailed explanations of the study in their native language.

Impact:

This study is expected to:

1. Enhance understanding of post-TB sequelae.
2. Inform clinical guidelines for TB survivor care.
3. Contribute to policy frameworks for managing long-term TB outcomes in resource-limited settings.
4. Provide pediatric insights into TB's impact on growth and development. This detailed description provides a comprehensive overview of the study's rationale, objectives, methodology, and anticipated outcomes. Let me know if further elaboration or refinement is needed!

ELIGIBILITY:
Inclusion Criteria for TB exposed group:

1. Children and adolescents aged 6 months to 15 years; and participants aged >15 years and above.
2. Successful completion of anti-TB treatment for the first episode of pulmonary TB and or pleural TB, with cure or completion as defined by the NTP.
3. Residing within Dhaka city and be willing to come for follow-up visits.(21)
4. Provide consent for participation to the study.

Exclusion Criteria for TB exposed group:

1. Past TB disease or anti-TB treatment within last 6 months.
2. Tuberculous meningitis, and isolated other extra-pulmonary TB (i.e no concomitant pulmonary TB, or pleural TB), multidrug resistant TB.
3. Participants getting immunosuppressive therapy or other chemotherapy for malignancy.
4. Pre-existing mental illness. Participants with preexisting mental illness will be identified based on documented prescriptions or medical records provided by a qualified physician.
5. Participants with known congenital heart disease, ischemic heart disease, cystic fibrosis. These participants will be identified based on documented prescriptions or medical records provided by a qualified physician.
6. Heavy smoker who consumes more than 20 pieces of cigarettes per day or ≥20 more pack-year.

Inclusion Criteria of TB Unexposed group:

age and sex-matched participants who do not have exposure to TB to compare post-TB sequelae data of study TB patients with that of a local non-TB population.

Exclusion Criteria of TB Unexposed group:

*Patient will be excluded if any two symptoms or signs suggestive of TB is present according to the national guidelines for the management of TB in children and adult.

Past TB disease or anti-TB treatment Any current or past (chronic) respiratory infection or disease.

* Documented pneumonia, bronchiolitis, bronchitis in last 3 weeks.
* Documented asthma, COPD, heart failure diagnosed by medical personnel
* Documented general wheezing in chest (last 2 years)
* Self-reported breathing difficulties during mild exercise, or at night. Heavy smoker who consumes more than 20 pieces per day or ≥20 more pack-year.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited through icddr,b Tuberculosis Screening & Treatment Centers (TBSTC) in Dhaka, where TB patients were referred for diagnosis and treatment initiation. Participants will be enrolled from seven TBSTCs in Mohakhali, Golapbagh, Dhanmondi, Uttara, Rampura, Mirpur, and Old Dhaka. These centers are managed by icddr,b under the National Tuberculosis Program (NTP) of Bangladesh. Additionally, child TB cases will be enrolled from Dhaka Shishu Hospital and icddr,b's Dhaka Hospital. Screening will occur during participants' monthly medication collection visits, with formal recruitment at the end of their TB treatment. To compare post-TB sequelae, age and sex-matched participants without TB exposure will be recruited from the same or neighboring households of study TB patients to serve as controls, allowing comparison of post-TB outcomes with the local non-TB population.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Understanding the post-intervention TB sequelae in patients after completion of standard TB treatment | Participants is enrolled within 5-7 days of TB treatment completion (T0) and follow-up is done at five time points: at 6 months (T1), 12 months (T2), 18 months (T3), and 24 months (T4)
  The primary end point will be the prevalence of Post TB Lung Disease (PTLD) among young children, older children and adults. We will define Post TB sequelae or PTLD as evidence of one or more chronic respiratory abnormality attributable at least in part to previous PTB or pleural TB, such as, chronic cough (persistent cough that lasts ≥8 weeks on some or most days); dyspnoea using the modified Medical Research Council (mMRC) dyspnoea scale; hypoxaemia (SpO2 <90% in room air); abnormal lung function test, and abnormal radiology findings after completion of TB treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- icddrb Dhaka hospital, Nutrition research division, Dhaka, Dhaka Division, Bangladesh